CLINICAL TRIAL: NCT04112498
Title: A Phase 1, Multi-Tumor, Bioavailability Study of Relatlimab in Combination With Nivolumab
Brief Title: A Phase 1, Bioavailability Study of Relatlimab in Combination With Nivolumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA224-087
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nivolumab + relatlimab + rHuPH20 (Experimental)
  Interventions: Drug: relatlimab; Drug: nivolumab; Drug: rHuPH20

INTERVENTIONS:
Drug: relatlimab — Specified dose on Specified days
Drug: nivolumab — Specified dose on Specified days
  Other Names: Opdivo
Drug: rHuPH20 — Specified dose on Specified days
  Other Names: Enhanze

SUMMARY:
This study will characterize the movement of drugs within the body, evaluate safety and determine to which extent the body can process relatlimab in combination with nivolumab in subjects with certain advanced tumors

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologic or cytologic confirmation of (unresectable and/or metastatic) advanced solid tumors
* Melanoma
* Metastatic squamous or non- squamous non-small cell lung cancer (NSCLC)
* Gastric adenocarcinoma (includes gastro-esophageal junction)
* Hepatocellular carcinoma (HCC)
* Squamous cell carcinoma of the head and neck (SCCHN)
* Renal cell carcinoma (RCC)
* Bladder cancer
* Participants must have received available standard therapies
* Women and men must agree to follow instructions for method of contraception
* Measureable disease as per RECIST version 1.1 criteria
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Participants must not have active brain metastases or leptomeningeal metastases
* Participants with HCC must not have any history of hepatic encephalopathy, any prior (within 1 year) or current clinically significant ascites
* History of allergy or hypersensitivity to study drug components
* Participants with serious or uncontrolled cardiovascular disease
* Excluding patients with serious or uncontrolled medical disorders
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment
* Participants with an active, known, or suspected autoimmune disease
* Participants must not have evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population

Other protocol defined inclusion/exclusion Criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
maximum observed serum concentration (Cmax) | approximately 60 days
time of maximum observed serum concentration (Tmax) | approximately 60 days
area under the time-concentration curve over the dosing interval AUC (TAU) | approximately 60 days
Observed concentration at the end of the dosing interval (Ctau) | approximately 60 days
Incidence of Serious Adverse Events (SAEs) | approximately 2 years
Incidence of Adverse Events (AEs) | approximately 2 years
Incidence of Adverse Events leading to discontinuation | approximately 2 years
Number of deaths | approximately 2 years
Number of laboratory abnormalities | approximately 2 years

SECONDARY OUTCOMES:
Incidence of Adverese Events (AEs) in the broad SMQ of Anaphylactic Reaction | approximately 2 years
Number of events within the hypersensitivity/infusion reaction select AE category | approximately 2 years
Incidence of anti-relatlimab antibodies and neutralizing antibodies (if applicable) | approximately 2 years
Incidence of anti-nivolumab antibodies and neutralizing antibodies (if applicable) | approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution - 0001, Hackensack, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome